CLINICAL TRIAL: NCT07080749
Title: The Effects of Vagus Nerve Stimulation on Pain, Muscle Stiffness, Heart Rate, And Functional Activities in Individuals With Chronic Widespread Pain - A Double Blinded Randomized Control Trial
Brief Title: The Effect of Vagus Nerve Stimulation on Pain and Functional Activities in Individuals With Chronic Widespread Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Georgia (Other)
Responsible Party: Principal Investigator, Mohammad(Reza) Nourbakhsh, Professor of Physical Therapy, University of North Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Number 2025-048
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Widspread Chronic Pain, Fibromyalgia
Keywords: Vagal Nerve Stimulation; Deep Exhalation; Ear Electrical Stimulation; Chronic Pain; Central Sensitization
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Observation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vagal Nerve Stimulation through deep exhalation. (Active Comparator): Vagal nerve stimulation will be performed through deep exhalation exercise, performed once every hour during the waking hours each day.
  Interventions: Other: Vagal nerve stimulation through deep exhalation exercise
- Vagal Nerve Stimulation through ear electrical stimulation (Active Comparator): Vagal nerve stimulation will be performed through applying low frequency electrical stimulation to the external ear lobe for 20 minutes twice a day.
  Interventions: Other: Vagal nerve stimulation through ear electrical stimulation
- No intervention (Other): Participants in this group will not receive any treatment for vagal nerve stimulation.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: Vagal nerve stimulation through deep exhalation exercise — Deep Exhalation Treatment: Participants will receive a set of standard balloons to use for deep exhalation. They will sit in a comfortable position, take a deep breath in and blow their breath continuously out into the balloon. They repeat the deep exhalation process for a total of 4 consecutive breaths. They perform this breathing exercise once every hour during waking hours each day.
  Arms: Vagal Nerve Stimulation through deep exhalation.
Other: Vagal nerve stimulation through ear electrical stimulation — Ear Electrical Stimulation Treatment: Participants will receive a small electrical stimulator and electrode set to be applied to their left ear. The investigators will train the participants to use the device safely and effectively. Once they are comfortable with the procedure, they will perform the procedure at home for 20 minutes twice daily.
  Arms: Vagal Nerve Stimulation through ear electrical stimulation
Other: No intervention (observational study) — The no intervention group will not receive treatment immediately after their baseline assessments, they will be scheduled for another visit after two weeks, then a new set of baseline measurements will be recorded as the post intervention data.
  Arms: No intervention

SUMMARY:
The goal of this clinical trial is to examine the effect of vagus nerve stimulation (VNS) on chronic, widespread pain in adults. The study will also evaluate which method of VNS-electrical ear stimulation or deep exhalation breathing-has a more significant impact on pain intensity, quality of life, and emotional well-being.

The main questions it aims to answer are:

Does vagus nerve stimulation reduce pain intensity in individuals with chronic, widespread pain?

Which intervention-electrical ear stimulation or deep exhalation breathing-provides a greater improvement in autonomic function, emotional status, and quality of life?

Researchers will compare two active interventions-electrical ear stimulation and deep exhalation breathing-to a no-treatment control group to determine relative effectiveness on pain and related outcomes.

Participants will:

Be randomly assigned to one of three groups:

* Electrical Ear Stimulation: Apply a small, non-invasive device to the ear for 20 minutes, twice daily for two weeks.
* Deep Exhalation Breathing: Perform balloon-blowing exercises (four deep exhalations per set) once every waking hour each day for two weeks.
* Control Group: Receive no intervention during the two-week period. These participants will complete baseline testing, return after two weeks for follow-up testing, and then be debriefed. They will have the option to withdraw or receive an active treatment after study data collection concludes.

Complete four questionnaires to assess pain, emotional state, and quality of life.

Undergo physiological assessments including heart rate variability, neck muscle tissue flexibility (via MyotonPro), and pressure pain sensitivity (via pressure algometer), both before and after the 2-week period.

Participation includes two in-person sessions (approximately 1 hour each) and daily home practice (for intervention groups) lasting 40-60 minutes per day for two weeks. The study involves minimal risk, and no compensation is provided. Participation is voluntary, and confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
Detailed Description:

Study Overview:

This randomized controlled clinical trial investigates the effects of two forms of non-invasive vagus nerve stimulation (VNS) on chronic widespread pain (CWP). The study is designed to explore whether stimulating the vagus nerve through auricular electrical stimulation (AES) or deep forced exhalation (DFE) improves pain, muscle stiffness, and functional status in individuals with CWP.

Vagal nerve stimulation (VNS) has been associated with modulation of the autonomic nervous system, leading to downstream effects on inflammation, pain perception, and emotional regulation. This study compares the effectiveness of these two intervention methods with a control group that receives no treatment during the study period.

Research Questions:

1. Does VNS via deep forced exhalation improve pain, muscle stiffness, and functional outcomes in individuals with chronic widespread pain?
2. Does VNS via auricular electrical stimulation improve these same outcomes?
3. Is one intervention more effective than the other in improving autonomic and pain-related parameters?

Hypotheses:

* Null Hypothesis: Neither deep forced exhalation nor auricular electrical stimulation will produce significant improvements in pain, muscle stiffness, or functional capacity.
* Alternative Hypothesis: Both interventions will lead to significant improvements in pain, muscle stiffness, and functional outcomes compared to a control group.

Study Procedures and Assessments:

Participants will be randomly assigned to one of three groups:

1. Auricular Electrical Stimulation (AES)
2. Deep Forced Exhalation (DFE)
3. No-Treatment Control Each participant will undergo the same battery of assessments at baseline and after the two-week intervention or observation period.

<!-- -->

1. Heart Rate Variability (HRV):

   Assessed using the Polar H10 chest strap sensor.
   * Equipment preparation: The investigator ensures the Polar H10 sensor and strap are clean and functional. Electrode areas are moistened with water or gel to improve signal quality. Bluetooth is enabled on the recording device (e.g., smartphone).
   * Participant setup: Participants wear clothing allowing chest access. The chest strap is positioned snugly around the torso, just below the chest muscles and centered on the sternum. The Polar H10 sensor is connected to the chest strap for data collection. and ensure it activates (indicated by a blinking LED light).
   * Data collection: The participant sits in a relaxed upright posture in a quiet, temperature-controlled room. After a 5-minute acclimation period, HRV data is recorded for 10 minutes. Participants are instructed not to talk, move, or use electronic devices during this time.
2. Muscle Stiffness and Tissue Compliance:

   Measured using the MyotonPRO device on the upper trapezius. • Equipment preparation: The MyotonPRO is calibrated before each session.

   • Participant setup: The participant wears clothing that allows shoulder access and avoids caffeine, alcohol, or vigorous activity for at least 2 hours prior. The participant lies supine for at least 5 minutes before testing.

   • Measurement: The skin is cleaned and the midpoint of the trapezius marked. The probe is placed perpendicular to the skin, and 3-5 consecutive measurements are taken on each side. The device records stiffness (N/m), elasticity, relaxation time, frequency, and compliance. Data is stored under a participant ID for analysis.
3. Pain Pressure Threshold (PPT):

   Assessed with a handheld analog pressure algometer at three locations: mid trapezius, L5 lumbar paraspinal, and gastrocnemius-soleus junction.
   * Setup: The participant avoids caffeine, alcohol, and intense activity for at least 2-3 hours. They rest for 5-10 minutes in a quiet room before testing.
   * Protocol: Skin is marked, and the procedure is explained. Pressure is applied at ~30 kPa/sec until the participant signals when it transitions to pain. Three trials are performed at each site with 30-60 second rests. The average of three values is recorded.
4. Pain Level:

   Measured using the Visual Analog Scale (VAS), a 10 cm line from "no pain" to "worst pain imaginable."
5. Quality of Life:

   Measured with the Quality of Life Scale (QOLS), covering physical, emotional, and social domains.
6. Emotional State:

   Assessed using the Positive and Negative Affect Schedule (PANAS), which rates 10 positive and 10 negative emotions.
7. Depression Severity:

Evaluated using the Patient Health Questionnaire-9 (PHQ-9), a 9-item tool commonly used in research and clinical practice.

Intervention Protocols:

1. Auricular Electrical Stimulation (AES):

   • Objective: Stimulate the auricular branch of the vagus nerve (ABVN) using taVNS.

   • Site: Cymba conchae of the left ear.

   • Equipment: Standard taVNS device, clip electrodes with conductive gel, timer, and alcohol swabs.

   • Stimulation Parameters:

   o Waveform: Biphasic rectangular

   o Pulse width: 200-300 µs

   o Frequency: 20 Hz

   o Intensity: Starting at 0.1 mA, increased until tingling is comfortable but not painful

   o Duration: 20 minutes per session, twice daily for 2 weeks

   • Contraindications: Cardiac arrhythmia, implanted pacemakers, pregnancy, epilepsy, skin infection at site, metal implants near ear.
   * Procedure: First session is supervised. Participants are trained to apply the device at home. Instructions emphasize safety, comfort, and proper use. Participants remain seated or semi-reclined during stimulation, and are instructed to avoid standing or walking while stimulated.
2. Deep Forced Exhalation (DFE):

   • Objective: Stimulate vagal tone through autonomic regulation via breathwork.
   * Equipment: Latex-free balloons and logbook.
   * Procedure: Participants take a deep breath, blow continuously into the balloon, then block airflow with the tongue. This is repeated for 4 breaths. The procedure is practiced once per hour during waking hours. Participants sit comfortably and avoid physical strain.
3. Control Group:

Participants undergo all pre- and post-study assessments but receive no intervention during the two-week period. They are debriefed afterward and may opt to receive either treatment following data collection.

Safety Considerations:

Potential AES risks include local irritation, tingling, warmth, lightheadedness, or bradycardia. All participants are screened and monitored during the first session. Instructions emphasize safe positioning, hydration, and gradual adjustment of intensity. Participants are advised to stop the session and contact the research team if they feel unwell.

DFE carries low risk, with occasional lightheadedness or fatigue reported. This is minimized by recommending seated practice and gradual breath intensity. Participants are asked to rest after each session.

Expected Benefits:

Participants may experience decreased pain sensitivity, improved autonomic regulation, better emotional well-being, and improved quality of life. These outcomes are not guaranteed, and no monetary compensation is offered for participation.

Contact Information:

Dr. Reza Nourbakhsh Email: Reza.nourbakhsh@ung.edu Phone: 706-864-1766

ELIGIBILITY:
Inclusion Criteria:

Adults 18 years of age or older

Diagnosed by a healthcare provider with chronic widespread pain or fibromyalgia

Exclusion Criteria:

Cardiovascular disorders: Such as arrhythmia (irregular heartbeat), heart failure, coronary artery disease, or history of heart surgery

Neurological disorders: Including epilepsy, Parkinson's disease, multiple sclerosis, neuropathy, or seizures

Endocrine disorders: Such as uncontrolled diabetes, thyroid disease (hypothyroidism or hyperthyroidism), or adrenal disorders

Gastrointestinal disorders: Including inflammatory bowel disease (Crohn's disease, ulcerative colitis), irritable bowel syndrome, or chronic acid reflux (GERD)

Respiratory disorders: Such as asthma, chronic bronchitis, emphysema, or sleep apnea

Vestibular disorders: Including Meniere's disease, benign paroxysmal positional vertigo (BPPV), or any condition causing balance problems

History of concussion or traumatic brain injury

Frequent dizziness or vertigo: History of unexplained or recurring episodes

Chronic or recurrent headaches: Including migraines, tension-type headaches, or cluster headaches

Ear problems: History of ear infections, hearing loss, tinnitus (ringing in the ears), or ear surgeries

Throat problems: History of chronic sore throat, difficulty swallowing (dysphagia), or throat surgery

Herniation: History of any type of herniation such as spinal disc herniation, inguinal (groin) hernia, or abdominal hernia

Skin sensitivity to electrical stimulation: Known allergic reaction, rash, or irritation from electrode pads or electrical devices applied to the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From enrollment to the end of treatment at 2 weeks
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10 cm horizontal line anchored by "no pain" and "worst imaginable pain." Participants mark their current level of pain on the line, which is measured in centimeters (cm).
Muscle stiffness | Frome enrollment to the end of treatment at 8 weeks
  Muscle stiffness, defined as the resistance of the tissue to an external force, will be measured in the upper trapezius using the MyotonPro device. Stiffness reflects the biomechanical integrity of muscle tissue. Unit of Measure: Newtons per meter (N/m)
Pressure Pain Threshold - Trapezius muscle | From enrollment to the end of treatment period at 2 weeks
  Pressure pain threshold (PPT) at the mid-belly of the upper trapezius will be assessed using a calibrated analog pressure algometer. PPT is defined as the minimum force required to elicit pain and reflects mechanical pain sensitivity. Unit of Measure: Kilograms per square centimeter (kg/cm²).
SDNN (Standard Deviation of NN intervals) | From enrollment to the end of treatment at 2 weeks
  SDNN will be used to assess overall heart rate variability, reflecting both sympathetic and parasympathetic nervous system activity over a 10-minute resting period. Unit of Measure: milliseconds (ms).
Mechanical Stress Relaxation Time | From enrollment to the end of treatment at 8 weeks
  Mechanical Stress Relaxation Time, defined as the time required for tissue to return to its original state following a mechanical impulse, will be measured using the MyotonPro device. This parameter reflects the viscoelastic properties of skeletal muscle. Unit of Measure: milliseconds (ms).
Muscle Oscillation Frequency | From enrollment to the end of treatment at 8 weeks.
  Frequency, representing the natural oscillation frequency of muscle tissue in response to a brief mechanical impulse, will be measured using the MyotonPro device. It reflects the intrinsic muscle tone and biomechanical behavior of the tissue. Unit of Measure: Hertz (Hz).
Pressure Pain Threshold - Lumbar Paraspinal Muscles | From enrollment to the end of treatment at 8 weeks
  PPT at the lumbar paraspinal region (L5 level) will be measured using an analog pressure algometer to assess localized pain sensitivity. Unit of measurement: Kilograms per square centimeter (kg/cm²)
Pressure Pain Threshold - Calf Muscles | From enrollment to the end of treatment at 8 weeks
  PPT at the junction of the gastrocnemius and soleus muscles in the calf will be measured using a pressure algometer to evaluate distal pain sensitivity. Unit of Measure: Kilograms per square centimeter (kg/cm²)
Muscle Elasticity (Logarithmic Decrement) | From enrollment to the end of treatment at 8 weeks
  Elasticity, measured as logarithmic decrement, describes the ability of muscle tissue to return to its original shape after deformation. It will be measured using the MyotonPro on the upper trapezius. Lower values indicate greater elasticity. Unit of Measure: Unitless (logarithmic decrement)
RMSSD (Root Mean Square of Successive Differences) | Baseline, after 2 weeks and after 8 weeks
  RMSSD will be used as a marker of short-term parasympathetic activity. Unit of Measure: milliseconds (ms).
SDANN (Standard Deviation of Average NN intervals) | Baseline, after 2 weeks, and after 8 weeks
  SDANN will be used to evaluate longer-term components of heart rate variability associated with sympathetic activity. Unit of Measure: milliseconds (ms)
LF Power (Low Frequency Power) | Baseline, after 2 weeks and after 8 weeks
  LF Power will be analyzed to assess contributions from both sympathetic and parasympathetic nervous systems in frequency domain. Unit of Measure: milliseconds² (ms²).
HF Power (High Frequency Power) | Baseline, after 2 weeks and after 8 weeks
  HF Power will be measured to evaluate parasympathetic (vagal) nervous system activity. Unit of Measure: milliseconds² (ms²).
LF/HF Ratio | Baseline, after 2 weeks and after 8 weeks
  LF/HF ratio will be used as a marker of autonomic balance, indicating the relative influence of sympathetic to parasympathetic tone. Unit of Measure: Ratio (unitless).
VLF Power (Very Low Frequency Power) | Baseline, after 2 weeks and after 8 weeks
  VLF Power will be measured to assess longer-term regulatory systems, including thermoregulation and hormonal factors. Unit of Measure: milliseconds² (ms²).
ULF Power (Ultra Low Frequency Power) | Baseline, after 2 weeks and after 8 weeks
  ULF Power will be assessed to capture circadian and ultradian influences on autonomic regulation. Unit of Measure: milliseconds² (ms²).

SECONDARY OUTCOMES:
Quality of Life (Quality of Life Scale - QOLS) | From enrollment to the end of treatment period at 2 weeks.
  The Quality of Life Scale (QOLS) will be used to evaluate participants' perceived well-being and life satisfaction across physical, social, and personal domains. The scale includes 16 items scored from 1 to 7, with total scores ranging from 16 to 112. Unit of Measure: Total score (range: 16-112). Higher scores indicate better quality of life.
Positive Affect Score (PANAS) | From enrollment to the end of treatment period at 2 weeks
  The Positive and Negative Affect Schedule (PANAS) will be used to assess emotional state. The positive affect subscale contains 10 items, each rated from 1 (very slightly or not at all) to 5 (extremely), yielding scores from 10 to 50. Unit of Measure: Total score (range: 10-50). Higher scores indicate a higher level of positive emotional state.
Depression Severity (Patient Health Questionnaire-9) | From enrollment to the of treatment period at 2 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report scale measuring depression symptom severity. Each item is rated from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. Unit of Measure: Total score (range: 0-27). Higher scores indicate more severe depressive symptoms.
Negative Affect Score (Positive and Negative Affect Schedule - PANAS) | From enrollment to the end of treatment at 8 weeks
  The PANAS negative affect subscale consists of 10 items, each scored from 1 to 5, with a total score ranging from 10 to 50. This subscale measures levels of distress and negative emotionality. Unit of Measure: Total score (range: 10-50). Higher scores indicate greater negative emotional states.
Muscle Creep/Compliance | From enrollment to the end of treatment at 8 weeks
  Creep (or compliance), representing the viscoelastic behavior of muscle over time, will be assessed using the MyotonPro device. This parameter reflects the ability of muscle tissue to deform gradually under sustained stress. Unit of Measure: Deborah number (or dimensionless unit, based on device output)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Georgia, Dahlonega, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication with no end date
Access Criteria: A data sharing agreement must be signed